CLINICAL TRIAL: NCT01866358
Title: Intraosseous Infusion for Neonatal Asphyxiated Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Lixue, director，head nurse of pediatric department ，principal investigator ，clinical professor, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Wanglan
Record Dates: First submitted 2013-05-21; First posted 2013-05-31 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Asphyxia Neonatorum
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Infusions, Intraosseous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Umbilical vein infusion (Placebo Comparator): using umbilical vein infusion for resucitation
  Interventions: Procedure: Umbilical vein infusion
- Intraosseous infusion (Experimental): using intraosseous infusion for resucitation
  Interventions: Procedure: Intraosseous infusion

INTERVENTIONS:
Procedure: Intraosseous infusion — Using intraosseous infusion for resustation in this group
  Arms: Intraosseous infusion
Procedure: Umbilical vein infusion — Using umbilical vein infusion for resustation in this group
  Arms: Umbilical vein infusion

SUMMARY:
Intraosseous infusion is better than umbilical vein infusion for neonatal asphyxiated resuscitation

ELIGIBILITY:
Inclusion Criteria:

* newborns who need resucitation

Exclusion Criteria:

-

Ages: 28 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
success rate of resuscitation | 24 hours

SECONDARY OUTCOMES:
Injury of brain and heart | 1 month

OTHER OUTCOMES:
Success rate of puncture | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD, Study Chair — Professor, Chief of Pediatric Department
Locations (1):
- Pediatrics of Daping Hospital, Chongqing, Chongqing Municipality, China